CLINICAL TRIAL: NCT05723354
Title: Comparison of Clinical Efficacy of Axillary Block in Patients of Cervical Radiculopathy
Brief Title: Clinical Efficacy of Axillary Block in Cervical Radiculopathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Keimyung University Dongsan Medical Center (Other)
Responsible Party: Principal Investigator, Ji Hee Hong, Professor, Keimyung University Dongsan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023-01-025-05
Record Dates: First submitted 2023-02-03; First posted 2023-02-10 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Pain, Chronic
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 5ml axillary block group (Active Comparator): interfascial plane axillary block group using 5 ml local anesthetics
  Interventions: Procedure: axillary block guided by ultrasound
- 10ml axillary block group (Active Comparator): interfascial plane axillary block group using 10 ml local anesthetics
  Interventions: Procedure: axillary block guided by ultrasound

INTERVENTIONS:
Procedure: axillary block guided by ultrasound — axillary block using local anesthetics

SUMMARY:
The primary endpoint of this study was to compare the clinical efficacy of axillary block in patients of cervical radiculopathy using 2 volumes of local anesthetics.

DETAILED DESCRIPTION:
The interscalene brachial plexus block is an effective intervention for reducing postoperative pain but is related to side effects, Suprascapular nerve block and a block of the axillary nerve have been introduced as alternatives to the interscalene brachial plexus for the control of postoperative pain. Previous study demonstrated new method of axillary block using interfascial plane injection guided by ultrasoud. Axillary block has been used widely for the relief of postoperative arm pain.

Recent study deomonstrated good pain relief when ultrasound guided interfascial plane injection was performed in patients with cervical radiuculopathy.

There is no study showing clinical efficacy of interfascial plane injection of axillary block in patients of cervical radiculopathy.

ELIGIBILITY:
Inclusion Criteria:

* Cervical foraminal stenosis
* Cervical central stenosis
* Cervical disc herniation
* Cervical spondylolisthesis
* Prominent arm pain rather than neck pain

Exclusion Criteria:

* Infection
* Pregnancy
* allergy to local anesthetic agents
* previous cervical spine surgery
* Prominent neck pain rather than arm pain

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-02-13 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Numerical rating scale changes among 4 time periods | baseline, 2 weeks after injection, 4 weeks after injection, 8 weeks after injection
  Numerical rating scale changes among 4 time periods
Neck disability injex changes between 2 time periods | baseline, 8 weeks after injection
  Neck disability injex changes between 2 time periods

CONTACTS AND LOCATIONS:
Locations (1):
- Hong ji HEE, Daegu, South Korea